CLINICAL TRIAL: NCT01318824
Title: A Study of Bi-Level Positive Airway Pressure (BIPAP) Versus Non Invasive Positive Pressure Ventilation (NIPPV) for Neonatal Respiratory Failure
Acronym: BIPAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Yuan Shi and Shifang Tang, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011002
Record Dates: First submitted 2011-02-23; First posted 2011-03-21 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-01

CONDITIONS: Neonatal Respiratory Failure
Keywords: Neonatal Respiratory Failure; Newborn Infant; BiPAP; NIPPV

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I=NIPPV (Placebo Comparator): This group receiving Nasal Intermittent Positive Pressure Ventilation (NIPPV) treatment.
  Interventions: Procedure: Nasal Intermittent Positive Pressure Ventilation (NIPPV)
- II=BiPAP (Experimental): This group receive Bi-Level Positive Airway Pressure (BIPAP) treatment
  Interventions: Procedure: Bi-Level Positive Airway Pressure (BIPAP)

INTERVENTIONS:
Procedure: Nasal Intermittent Positive Pressure Ventilation (NIPPV) — The Control group receiving Nasal Intermittent Positive Pressure Ventilation (NIPPV) treatment
  Other Names: Nasal Intermittent Positive Pressure Ventilation
  Arms: I=NIPPV
Procedure: Bi-Level Positive Airway Pressure (BIPAP) — BiPAP group receive Bi-Level Positive Airway Pressure (BIPAP) treatment
  Other Names: Bi-Level Positive Airway Pressure
  Arms: II=BiPAP

SUMMARY:
To research the effect of Bi-Level Positive Airway Pressure (BiPAP) for neonatal respiratory failure.

DETAILED DESCRIPTION:
Bi-Level Positive Airway Pressure(BiPAP) is similar to Non Invasive Positive Pressure Ventilation (NIPPV), but also gives some breaths, or extra support, to newborn infants through a small tube in the nose. BiPAP is safe and effective. Nevertheless, BiPAP has never been used in Chinese babies.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn infants with birth weight > 500 gm.
2. Gestational age > 24 completed weeks.
3. Intention to manage the infant with non-invasive respiratory support (i.e. no endotracheal tube), where either: the infant is within the first 7 days of life and has never been intubated or has received less than 24 hours of total cumulative intubated respiratory support the infant is within the first 28 days of life, has been managed with intubated respiratory support for 24 hours or more and is a candidate for extubation followed by non-invasive respiratory support.
4. No known lethal congenital anomaly or genetic syndromes.
5. Signed parental informed consent.

Exclusion Criteria:

1. Considered non-viable by clinician (decision not to administer effective therapies)
2. Life-threatening congenital abnormalities including congenital heart disease (excluding patent ductus arteriosis)
3. Infants known to require surgical treatment
4. Abnormalities of the upper and lower airways
5. Neuromuscular disorders
6. Infants who are > 28 days old and continue to require mechanical ventilation with an endotracheal tube

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
the effect of Non Invasive Positive Pressure Ventilation (NIPPV) for Neonatal Respiratory Failure | At 7 days, 28 days and at 36 weeks postmenstraul age
  get the effect of Non Invasive Positive Pressure Ventilation (NIPPV) for Neonatal Respiratory Failure

SECONDARY OUTCOMES:
the effect of Versus Bi-Level Positive Airway Pressure (BIPAP) for Neonatal Respiratory Failure | At 7 days, 28 days and at 36 weeks postmenstraul age
  get the effect of Versus Bi-Level Positive Airway Pressure (BIPAP) for Neonatal Respiratory Failure

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, MD, Study Director — Department of Pediatrics, Daping Hospital, Third Military Medical University; Shifang Tang, Principal Investigator — Department of Pediatrics, Daping Hospital, Third Military Medical University
Locations (1):
- Deaprtment of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China